CLINICAL TRIAL: NCT05365204
Title: A Study for Optimization of 6% Hydroxyethyl Starch Based Indocyanine Green Near-infrared Fluorescence Navigated Sentinel Lymph Node Biopsy for Breast Cancer Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 111-009-F
Record Dates: First submitted 2022-04-27; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Sentinel Lymph Node
Keywords: Indocyanine green; Sentinel lymph node biopsy; Axillary lymph node dissection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The participants will be assigned to sentinel lymph node biopsies using different concentrations of voluven based indocyanine green. Estimated concentration grouping (ICG mg / Voluven mL): 2.5, 0.5, 0.25, 0.125, 0.0625. Planned recruiting at least 3 participants in each diluted concentration group. The dilution rate will advance if imaging quality is improving compared with the last concentration group. The study will be completed if the best imaging quality injection protocol is found.
Who Masked: Participant
Masking Description: The participant will know how many concentration ladders we have, but will not know the exact concentration used on him.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Voluven diluted indocyanine green (Experimental): This arm participants uses Voluven diluted ICG for sentinel lymph node mapping.
  Interventions: Procedure: Near infrared fluorescence navigated sentinel lymph node mapping
- Distilled-water diluted indocyanine green (Active Comparator): This arm participants uses Distilled-water diluted ICG for sentinel lymph node mapping.
  Interventions: Procedure: Near infrared fluorescence navigated sentinel lymph node mapping

INTERVENTIONS:
Procedure: Near infrared fluorescence navigated sentinel lymph node mapping — Patient will undergo sentinel lymph node biopsy with near infrared fluorescence navigation. The dosage of ICG will not exceed 2.5 mg in total, and the volume of the assigned solvent will not exceed 5 mL in total.

SUMMARY:
A study for dosage-image optimization of 6% hydroxyethyl starch diluted indocyanine green for near-infrared fluorescence navigated sentinel lymph node mapping for breast cancer patient.

DETAILED DESCRIPTION:
Pre-clinical experiment has shown using 6% hydroxyethyl starch (Voluven®) as a solvent, compared with pure water, can improve brightness of indocyanine green particles at the same concentration. Similar findings have been addressed using human serum albumin as a solvent for indocyanine green in previous studies, but there was no report using 6% hydroxyethyl starch as a solvent till now. This study aims for clinical translation and optimization of 6% hydroxyethyl starch diluted indocyanine green in breast cancer patients undergoing sentinel lymph node biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer, adults

Exclusion Criteria:

* Patient aged < 20 years old
* Primary lesion without indication of sentinel lymph node biopsy in current guidelines (Low-risk ductal carcinoma in situ or metastatic breast cancer)
* Patient who is allergic to primary tracers (including Tc99m and blue dye)
* Patient who is allergic to indocyanine green

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-04-07 (Estimated); Study Completion 2023-04-07 (Estimated)

PRIMARY OUTCOMES:
Signal-to-background ratio (SBR) | through study completion, an average of 1 year
  Evaluates the SBR of the near-infrared fluorescence between the retrieved sentinel lymph nodes and the background.
Penetration depth | through study completion, an average of 1 year
  Evaluates the depth of the deepest visualized subcutaneous lymphatics in the breast

SECONDARY OUTCOMES:
Sentinel lymph nodes pathology | through study completion, an average of 1 year
  The positivity and number of retrieved sentinel lymph nodes at definitive pathology report.
Time to total visualization of breast subcutaneous lymphatics | through study completion, an average of 1 year
  The time from injection of indocyanine green to total visualization of breast subcutaneous lymphatics

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Chun Hsieh, MD, Study Chair — National Taiwan University Hospital Hsin-Chu Branch
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch Biomedical Park Hospital, Zhubei, HsinChu County, Taiwan

REFERENCES:
- [Background] Mieog JS, Troyan SL, Hutteman M, Donohoe KJ, van der Vorst JR, Stockdale A, Liefers GJ, Choi HS, Gibbs-Strauss SL, Putter H, Gioux S, Kuppen PJ, Ashitate Y, Lowik CW, Smit VT, Oketokoun R, Ngo LH, van de Velde CJ, Frangioni JV, Vahrmeijer AL. Toward optimization of imaging system and lymphatic tracer for near-infrared fluorescent sentinel lymph node mapping in breast cancer. Ann Surg Oncol. 2011 Sep;18(9):2483-91. doi: 10.1245/s10434-011-1566-x. Epub 2011 Mar 1. PMID 21360250